CLINICAL TRIAL: NCT06311032
Title: Clinician Decision Making Regarding Surveillance for Low-risk Intraductal Papillary Mucinous Neoplasms of The Pancreas
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 22-01227
Record Dates: First submitted 2024-03-08; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Surgery Risk Assessment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Vignettes with Risk Stratification Tool: Physicians will be posed with a series of three clinical case vignettes. Each vignette describes an IPMN of varying severity, and the physician will be asked determine whether they would continue or discontinue clinical surveillance in each case. Participants in this arm will be provided a risk stratification tool (DART-1) when presented with their clinical case vignettes.
  The DART-1 is a 5-question tool which calculates the probability (%) of IPMNs without worrisome features or high-risk stigmata at diagnosis.
- Vignettes without Risk Stratification Tool: Physicians will be posed with a series of three clinical case vignettes. Each vignette describes an IPMN of varying severity, and the physician will be asked determine whether they would continue or discontinue clinical surveillance in each case. Participants in this arm will be not be provided a risk stratification tool when presented with their clinical case vignettes.

SUMMARY:
The main objective of this study is to determine how physicians make decisions regarding surveillance of Intraductal Papillary Mucinous Neoplasm's (IPMN) of the pancreas.

DETAILED DESCRIPTION:
The study will employ a survey design that poses physicians with a series of three clinical case vignettes. Each vignette describes an IPMN of varying severity, and the physician will be asked determine whether they would continue or discontinue clinical surveillance in each case.

This will be a double-blinded randomized survey study, featuring two arms. Providers will be randomized to either be provided with, or not provided with a risk stratification tool (DART-1) when presented with their clinical case vignettes.

ELIGIBILITY:
Inclusion Criteria:

* Membership in either the PACYFIC or PRECEDE consortiums
* Physician with expertise in the management of IPMN
* Able and willing to complete survey

Exclusion Criteria:

* Not a member of either the PACYFIC or PRECEDE consortiums
* Not a physician with expertise in the management of IPMN

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The Pancreatic Cancer Early Detection (PRECEDE) Consortium is an international, multi-institutional collaborative group of experts to increase survival for pancreatic cancer patients by improving early detection, screening, risk modeling and prevention for those with a heritable risk for pancreatic cancer, through a novel model of collaboration and data sharing.
  The PACYFIC group is comprised of Dutch surgeons, gastroenterologists, oncologists, radiologists, radiotherapists, and pathologists. Their common interest is to improve the prognosis of patients with pancreatic cancer, by initiating and performing research, and organizing ongoing training.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2023-03-29 (Actual); Primary Completion 2023-06-28 (Actual); Study Completion 2023-07-28 (Actual)

PRIMARY OUTCOMES:
Number of Decisions to Stop Surveillance Imaging | Day 1
Number of Decisions to Continue Surveillance Imaging | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Greg Sacks, MD, MPH, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: Greg.Sacks@nyulangone.org. The statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to Greg.Sacks@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.